CLINICAL TRIAL: NCT06616818
Title: DASH Diet Intervention for Systemic Hypertension in Adolescents
Acronym: DISH
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding not awarded
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Carissa Baker-Smith, Professor of Pediatrics, Nemours Children's Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Nemours DASH Diet Study
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2024-09

CONDITIONS: Hypertension; Food Insecurity
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: 6 months of produce delivery.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- STANDARD (Placebo Comparator): Nutrition counseling only as part of standard of care
  Interventions: Other: nutrition counselling only
- DASH diet toolkit arm (Active Comparator): A group of participants receiving DASH diet intervention
  Interventions: Other: DASH-FV

INTERVENTIONS:
Other: DASH-FV — 12weeks of fruit and vegetable delivery to the home
  Arms: DASH diet toolkit arm
Other: nutrition counselling only — nutrition counselling as part of standard of care
  Arms: STANDARD

SUMMARY:
Parallel randomized clinical trial comparing DASH produce home delivery to routine care for the management of elevated blood pressure and hypertension in adolescents.

DETAILED DESCRIPTION:
Parallel randomized clinical trial comparing DASH produce home delivery to routine care for the management of elevated blood pressure and hypertension in adolescents.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 to 17 years of age at baseline visit
* Elevated blood pressure or hypertension

Exclusion Criteria:

* Inability to eat by mouth
* Secondary hypertension

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2026-08-01 (Estimated); Primary Completion 2031-08-31 (Estimated); Study Completion 2031-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in vegetable and fruit intake | 12 weeks and 6months
  Change in the average number of servings of vegetables and fruits consumed in a day.

SECONDARY OUTCOMES:
Systolic blood pressure | 12 weeks and 6 months
  Change in manual, in office systolic blood pressure

CONTACTS AND LOCATIONS:
Locations (1):
- Nemours Cardiac Center, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon request and upon completion.
Supporting Information: CSR
Time Frame: 6 months following study completion.
Access Criteria: Available upon request, but only deidentifed data.